CLINICAL TRIAL: NCT01499355
Title: A Multicenter, Randomized, Double-Blind, Placebo-Controlled Study to Evaluate the Efficacy, Safety, and Tolerability of BIIB023 in Subjects With Lupus Nephritis
Brief Title: BIIB023 Proof-of-Concept Study in Participants With Lupus Nephritis
Acronym: ATLAS
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Results from pre-specified criteria did not demonstrate sufficient efficacy to warrant continuation of the study.
Sponsor: Biogen (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 211LE201; 2011-002159-32 (EudraCT Number)
Record Dates: First submitted 2011-11-23; First posted 2011-12-26 (Estimated); Results first posted 2017-01-18 (Estimated); Last update posted 2017-01-18 (Estimated); Status verified 2016-11

CONDITIONS: Lupus Nephritis
MeSH Terms: conditions — Lupus Nephritis | interventions — BIIB023; Mycophenolic Acid; Adrenal Cortex Hormones

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Placebo (Placebo Comparator): Placebo intravenous (IV) infusion on Day 1, Week 2, Week 4, Week 8, and every 4 weeks thereafter through Week 48, plus background therapy including oral steroids (prednisone or equivalent) and mycophenolate mofetil (MMF)
  Interventions: Biological: Placebo; Drug: mycophenolate mofetil; Drug: oral corticosteroids
- BIIB023 3 mg/kg (Experimental): BIIB023 3 mg/kg IV on Day 1, Week 2, Week 4, Week 8, and every 4 weeks thereafter through Week 48 plus background therapy including oral steroids (prednisone or equivalent) and MMF.
  Interventions: Biological: BIIB023; Drug: mycophenolate mofetil; Drug: oral corticosteroids
- BIIB023 20 mg/kg (Experimental): BIIB023 20 mg/kg IV on Day 1, Week 2, Week 4, Week 8, and every 4 weeks thereafter through Week 48 plus background therapy including oral steroids (prednisone or equivalent) and MMF.
  Interventions: Biological: BIIB023; Drug: mycophenolate mofetil; Drug: oral corticosteroids

INTERVENTIONS:
Biological: BIIB023
  Arms: BIIB023 20 mg/kg; BIIB023 3 mg/kg
Biological: Placebo
  Arms: Placebo
Drug: mycophenolate mofetil — titrated to a target daily dose of 2 g (1 g twice daily)
  Other Names: MMF, Cellcept
Drug: oral corticosteroids — oral corticosteroids (prednisone or equivalent) at a target prednisone dose of 10 mg/day

SUMMARY:
The primary objective of the study is to assess the efficacy of BIIB023 as an add-on treatment to background therapy compared with placebo in combination with background therapy in the treatment of participants with active, biopsy-proven lupus nephritis. The secondary objectives of this study are to assess the safety and tolerability of BIIB023 compared with placebo in this study population.

DETAILED DESCRIPTION:
Participants who complete this study through Week 52 will be offered the option to enter an Extension study under a separate protocol 211LE202 (NCT0193089).

ELIGIBILITY:
Key Inclusion Criteria:

* Documented diagnosis of systemic lupus erythematosus (SLE) according to current American College of Rheumatology (ACR) criteria. At least 4 ACR criteria must be documented, 1 of which must be a positive antinuclear antibody (ANA), anti Sm, or anti dsDNA antibody.
* Diagnosis of International Society of Nephrology/Renal Pathology Society (ISN/RPS) 2003 Class III or IV lupus nephritis with either active or active/chronic disease, confirmed by biopsy within 3 months prior to Screening. Participants are permitted to have co existing Class V lupus nephritis. If a renal biopsy has not been performed within 3 months of the Screening Visit, one can be performed during the Screening Period after all other eligibility criteria have been confirmed. The local histological diagnosis must be confirmed by the central study pathologist.
* Must have proteinuria at Screening (from a 24 hour urine sample collection) defined as urinary protein:creatinine ratio (uPCR) >1.0 mg/mg.

Key Exclusion Criteria:

* Retinitis, poorly-controlled seizure disorder, acute confusional state, myelitis, stroke or stroke syndrome, cerebellar ataxia, or dementia that is currently active and resulting from SLE at Screening
* Estimated glomerular filtration rate (eGFR) <30 mL/min per 1.73 m^2 (calculated using the abbreviated Modification of Diet in Renal Disease equation) or the presence of oliguria or end-stage renal disease requiring dialysis or transplantation
* Subjects requiring dialysis within 12 months prior to Screening
* History of renal transplant
* Treatment with any biologic B-cell-depleting therapy (e.g., anti-CD20 [rituximab], anti-CD22 [epratuzumab], anti-BLyS/B-cell activating factor [e.g., briobacept, belimumab] therapy), or TACI-Ig within 12 months prior to Run-in Day 1.

NOTE: Other protocol defined Inclusion/Exclusion criteria may apply.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 276 (Actual)
Dates: Start 2012-07; Primary Completion 2015-12 (Actual); Study Completion 2015-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Biogen
Locations (57):
- United States (9):
  - Research Site, Torrance, California
  - Research Site, Orlando, Florida
  - Research Site, Boston, Massachusetts
  - Research Site, Rochester, Minnesota
  - Research Site, Lake Success, New York
  - Research Site, Chapel Hill, North Carolina
  - Research Site, Columbus, Ohio
  - Research Site, Memphis, Tennessee
  - Research Site, El Paso, Texas
- Argentina (7):
  - Research Site, Capital Federal, Ciudad Autonoma Buenos Aires
  - Research Site, Córdoba, Córdoba Province
  - Research Site, San Miguel de Tucumán, Tucumán Province
  - Research Site, Ciudad Autonoma Buenos Aires
  - Research Site, La Plata
  - Research Site, San Juan
  - Research Site, San Miguel de Tucumán
- Research Site, Melbourne, Victoria, Australia
- Belgium (2):
  - Research Site, Leuven
  - Research Site, Liège
- Brazil (2):
  - Research Site, Cuiabá, Mato Grosso
  - Research Site, São Paulo, São Paulo
- Colombia (3):
  - Research Site, Barranquilla
  - Research Site, Bogotá
  - Research Site, Medellín
- France (3):
  - Research Site, Pessac, Gironde
  - Research Site, Lille, Nord
  - Research Site, Paris
- Research Site, Mainz, Germany
- Hong Kong (2):
  - Research Site, Hong Kong
  - Research Site, Shatin
- Hungary (2):
  - Research Site, Budapest
  - Research Site, Debrecen
- Research Site, Pisa, Italy
- Malaysia (6):
  - Research Site, Kuching, Sarawak
  - Research Site, Ipoh
  - Research Site, Kuala Lumpur
  - Research Site, Kuala Selangor
  - Research Site, Pulau Pinang
  - Research Site, Selangor Darul Ehsan
- Mexico (5):
  - Research Site, Saltillo, Coahuila
  - Research Site, Cuauhtémoc
  - Research Site, León
  - Research Site, Mexico City
  - Research Site, San Luis Potosí City
- Research Site, Lima, Peru
- Philippines (2):
  - Research Site, Manila
  - Research Site, Quezon City
- Poland (2):
  - Research Site, Lodz
  - Research Site, Wroclaw
- Research Site, Coimbra, Portugal
- Russia (2):
  - Research Site, Moscow
  - Research Site, Saint Petersburg
- South Korea (2):
  - Research Site, Busan
  - Research Site, Gyeonggi-do
- Research Site, Sagunto, Spain
- Thailand (2):
  - Research Site, Bangkoknoi, Bangkok
  - Research Site, Patumwan, Bangkok

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: A total of 276 participants were enrolled and 203 completed the run-in period and qualified for randomization; of these, 15 participants were not randomized.
Groups:
- Run-In Period: All Enrolled Participants: At Run-in Day 1, participants entering the study received oral corticosteroid (prednisone or equivalent) starting at 0.75 mg/kg/day (maximum allowed dose of 60 mg/day) for 2 weeks and subsequently tapered over an 8-week period to 10 mg/day by Run-in Week 10. Following confirmation of eligibility, subjects also received mycophenolate mofetil (MMF) starting at Run-in Day 1 at a total dose of 1 g/day and titrated to a target dose of 2 g/day by Run-in Week 2.
- Double-Blind Period: Placebo: Placebo intravenous (IV) infusion on Day 1, Week 2, Week 4, Week 8, and every 4 weeks thereafter through Week 48, plus background therapy of oral steroids (prednisone or equivalent) and MMF.
- Double-Blind Period: BIIB023 3 mg/kg: BIIB023 3 mg/kg IV on Day 1, Week 2, Week 4, Week 8, and every 4 weeks thereafter through Week 48, plus background therapy of oral steroids (prednisone or equivalent) and MMF.
- Double-Blind Period: BIIB023 20 mg/kg: BIIB023 20 mg/kg IV on Day 1, Week 2, Week 4, Week 8, and every 4 weeks thereafter through Week 48, plus background therapy of oral steroids (prednisone or equivalent) and MMF.
Period: Run-In Period
Arm/Group | Run-In Period: All Enrolled Participants | Double-Blind Period: Placebo | Double-Blind Period: BIIB023 3 mg/kg | Double-Blind Period: BIIB023 20 mg/kg
Started | 276 | 0 | 0 | 0
Completed | 245 | 0 | 0 | 0
Not Completed | 31 | 0 | 0 | 0
Not completed — Study Termination | 15 | 0 | 0 | 0
Not completed — Other | 3 | 0 | 0 | 0
Not completed — Death | 2 | 0 | 0 | 0
Not completed — Investigator Decision | 2 | 0 | 0 | 0
Not completed — Consent Withdrawn | 1 | 0 | 0 | 0
Not completed — Adverse Event | 8 | 0 | 0 | 0
Period: Double-Blind Period
Arm/Group | Run-In Period: All Enrolled Participants | Double-Blind Period: Placebo | Double-Blind Period: BIIB023 3 mg/kg | Double-Blind Period: BIIB023 20 mg/kg
Started | 0 | 63 | 63 | 62
Completed | 0 | 40 | 38 | 39
Not Completed | 0 | 23 | 25 | 23
Not completed — Adverse Event | 0 | 2 | 3 | 2
Not completed — Study Termination | 0 | 18 | 16 | 14
Not completed — Other | 0 | 1 | 2 | 2
Not completed — Death | 0 | 1 | 0 | 0
Not completed — Investigator Decision | 0 | 0 | 3 | 3
Not completed — Consent Withdrawn | 0 | 0 | 1 | 2
Not completed — Lost to Follow-up | 0 | 1 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- All Enrolled Participants: At Run-in Day 1, participants entering the study received oral corticosteroid (prednisone or equivalent) starting at 0.75 mg/kg/day (maximum allowed dose of 60 mg/day) for 2 weeks and subsequently tapered over an 8-week period to 10 mg/day by Run-in Week 10. Following confirmation of eligibility, subjects also received MMF starting at Run-in Day 1 at a total dose of 1 g/day and titrated to a target dose of 2 g/day by Run-in Week 2.
Arm/Group | All Enrolled Participants
Number analyzed (Participants) | 276
Age, Continuous [Mean (Standard Deviation); unit: years] | 32.3 (10.11)
Gender [Count of Participants; unit: Participants]
  Female | 242
  Male | 34

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants Who Achieve a Complete or Partial Renal Response at Week 52
Description: Complete renal response is defined as: (1) urinary protein:creatinine ratio (uPCR) < 0.5 mg/mg with ≥ 50% reduction of uPCR from Day 1 (Baseline; from a 24 hour urine collection); and (2) estimated glomerular filtration rate (eGFR) within normal range. Partial renal response is defined as: (1) ≥ 50% reduction in uPCR from Day 1 (Baseline; from a 24-hour urine collection) and, (2) with one of the following: (a) uPCR of < 1.0 mg/mg if the Day 1 (Baseline) was ≤ 3.0 mg/mg, or, (b) uPCR < 3.0 mg/mg if the Day 1 (Baseline) ratio was > 3.0 mg/mg; and stabilization of renal function (eGFR + or - 25% of Day 1 [Baseline] or serum creatinine within normal range).
Time Frame: Week 52
Population: Participants in the modified intent-to-treat (mITT) population (participants in ITT population except for those who withdrew from study due to study early termination. Includes participants who completed Week 44 infusion and Visits at Week 52/Early Withdrawal and Week 56/End of Study but withdrew due to study early termination.)
Measure: Number (90% Confidence Interval); unit: percentage of participants
Groups:
- Placebo: Placebo IV infusion on Day 1, Week 2, Week 4, Week 8, and every 4 weeks thereafter through Week 48, plus background therapy including oral steroids (prednisone or equivalent) and MMF.
Arm/Group | Placebo | BIIB023 3 mg/kg | BIIB023 20 mg/kg
Number analyzed (Participants) | 48 | 49 | 48
percentage of participants | 25 [14.7 to 35.3] | 16 [7.6 to 25.0] | 31 [20.3 to 42.3]

2. Secondary Outcome: Percentage of Participants Who Achieve Complete Renal Response at Week 52
Description: Complete renal response is defined as uPCR < 0.5 mg/mg with ≥ 50% reduction of uPCR from Baseline (from a 24-hour urine collection) and eGFR within normal range.
Time Frame: Week 52
Population: Participants in the mITT population (participants in ITT population except for those who withdrew from study due to study early termination. Includes participants who completed Week 44 infusion and Visits at Week 52/early withdrawal and Week 56/End of Study but withdrew due to study early termination.)
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | BIIB023 3 mg/kg | BIIB023 20 mg/kg
Number analyzed (Participants) | 48 | 49 | 48
percentage of participants | 6 | 8 | 8

3. Secondary Outcome: Duration of Renal Response in Participants Who Achieve Complete Renal Response at Week 52
Description: Duration of response was calculated as the days in between the date of Week 52 visit and the date when the participant last became complete renal responder on or before Week 52 visit. Complete renal response: (1) uPCR <0.5 mg/mg with ≥ 50% reduction of uPCR from Day 1 (Baseline) (from a 24 hour urine collection); and (2) eGFR within normal range.
Time Frame: Week 52
Population: Participants in the mITT population (participants in ITT population except for those who withdrew from study due to study early termination. (Includes participants who completed Week 44 infusion and Visits at Week 52/Early Withdrawal and Week 56/End of Study but withdrew due to study early termination.)
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | BIIB023 3 mg/kg | BIIB023 20 mg/kg
Number analyzed (Participants) | 48 | 49 | 48
Participants
  1-day duration | 2 | 3 | 2
  27-day duration | 0 | 0 | 1
  78-day duration | 0 | 1 | 0
  141-day duration | 1 | 0 | 0
  169-day duration | 0 | 0 | 1

4. Secondary Outcome: Time to Renal Response (Partial or Complete) in Participants Who Achieve Renal Response at Week 52
Description: Onset of renal response was calculated as weeks elapsed from baseline date to first visit where renal response was achieved. Complete renal response is defined as: (1) uPCR <0.5 mg/mg with ≥ 50% reduction of uPCR from Day 1 (Baseline) (from a 24 hour urine collection); and (2) eGFR within normal range. Partial renal response is defined as: (1) ≥ 50% reduction in uPCR from Day 1 (Baseline; from a 24-hour urine collection) and, (2) with one of the following: (a) uPCR of < 1.0 mg/mg if the Day 1 (Baseline) was ≤ 3.0 mg/mg, or, (b) uPCR < 3.0 mg/mg if the Day 1 (Baseline) ratio was > 3.0 mg/mg; and stabilization of renal function (eGFR + or - 25% of Day 1 [Baseline] or serum creatinine within normal range). Estimated from the Kaplan-Meier Curve.
Time Frame: Baseline to Week 52
Population: Participants in the ITT population who achieved a renal response at Week 52. The ITT population included all participants who were randomized and received at least 1 dose of study treatment (BIIB023 or placebo).
Measure: Median (Full Range); unit: weeks
Arm/Group | Placebo | BIIB023 3 mg/kg | BIIB023 20 mg/kg
Number analyzed (Participants) | 12 | 8 | 15
weeks | 10.6 [2 to 41] | 5.2 [2 to 28] | 4.1 [2 to 37]
Statistical Analysis 1: Comparison: Placebo vs BIIB023 3 mg/kg; Test type: Superiority or Other; p = 0.367, Cox proportional hazard — P-Value from Cox proportional hazard model, including the variable for treatment, adjusted for the covariates including region (Latin America, Asia, rest of world [ROW]) and renal response at Run-in Week 12 (partial and non-response)
Statistical Analysis 2: Comparison: Placebo vs BIIB023 20 mg/kg; Test type: Superiority or Other; p = 0.283, Cox proportional hazard — P-Value from Cox proportional hazard model, including the variable for treatment, adjusted for the covariates including region (Latin America, Asia, ROW) and renal response at Run-in Week 12 (partial and non-response)

5. Secondary Outcome: Percentage of Participants With uPCR > 3.0 mg/mg at Baseline Who Achieve uPCR <1.0 mg/mg at Week 52
Time Frame: Baseline (Day 1), Week 52
Population: Participants with a uPCR > 3.0 mg/mg at Baseline in the mITT population (participants in ITT population except for those who withdrew from study due to study early termination. Includes those who completed Week 44 infusion and Visits at Week 52/Early Withdrawal and Week 56/End of Study but withdrew due to study early termination.)
Measure: Number (90% Confidence Interval); unit: percentage of participants
Arm/Group | Placebo | BIIB023 3 mg/kg | BIIB023 20 mg/kg
Number analyzed (Participants) | 12 | 18 | 15
percentage of participants | 0 [NA to NA] — No participants in this arm had a uPCR < 1.0 mg/mg at Week 52. | 22 [6.1 to 38.3] | 13 [0.0 to 27.8]
Statistical Analysis 1: Comparison: Placebo vs BIIB023 3 mg/kg; Test type: Superiority or Other; p = 0.0486, Cochran-Mantel-Haenszel — Model includes the variable for treatment, adjusted for the covariates including region (Latin America, Asia, ROW) and renal response at Run-in Week 12 (partial and non-response)
Statistical Analysis 2: Comparison: Placebo vs BIIB023 20 mg/kg; Test type: Superiority or Other; p = 0.0668, Cochran-Mantel-Haenszel — [p-value comment as in outcome 5, analysis 1]

6. Secondary Outcome: Percentage of Participants With Active Urinary Sediment at Baseline Who Have Inactive Urinary Sediment at Week 52
Description: Active urinary sediment is defined by 1 of the following (in the absence of a urinary tract infection or menses): > 5 red blood cell/high power field (RBC/HPF) or above the reference range for the laboratory, and > 5 white blood cell/high power field (WBC/HPF) or above the reference range for the laboratory, and presence of cellular casts (RBC or WBC). Inactive urinary sediment is defined as: < 5 RBC/HPF and < 5 WBC/HPF, or within the laboratory reference range, and no cellular casts (no RBC or WBC casts).
Time Frame: Baseline, Week 52
Population: Participants with active urinary sediment at Day 1 in the mITT population (participants in ITT population except for those who withdrew from study due to study early termination. (Includes participants who completed Week 44 infusion and Visits at Week 52/Early Withdrawal and Week 56/End of Study but withdrew due to study early termination.)
Measure: Number (90% Confidence Interval); unit: percentage of participants
Arm/Group | Placebo | BIIB023 3 mg/kg | BIIB023 20 mg/kg
Number analyzed (Participants) | 16 | 21 | 14
percentage of participants | 38 [17.6 to 57.4] | 5 [0.0 to 12.4] | 21 [3.4 to 39.5]
Statistical Analysis 1: Comparison: Placebo vs BIIB023 3 mg/kg; Test type: Superiority or Other; p = 0.0456, Regression, Logistic — [p-value comment as in outcome 5, analysis 1]; Odds Ratio (OR) = 0.0628, 90% CI 2-sided [0.0081 to 0.4843]
Statistical Analysis 2: Comparison: Placebo vs BIIB023 20 mg/kg; Test type: Superiority or Other; p = 0.5455, Regression, Logistic — [p-value comment as in outcome 5, analysis 1]; Odds Ratio (OR) = 0.4344, 90% CI 2-sided [0.0996 to 1.8941]
Statistical Analysis 3: Comparison: Placebo vs BIIB023 3 mg/kg; Test type: Superiority or Other; p = 0.0252, Cochran-Mantel-Haenszel
Statistical Analysis 4: Comparison: Placebo vs BIIB023 20 mg/kg; Test type: Superiority or Other; p = 0.2876, Cochran-Mantel-Haenszel

7. Secondary Outcome: Number of Participants With Adverse Events (AEs), Serious Adverse Events (SAEs) and AEs Leading to Study Discontinuation During the Run-In Period
Description: AEs that had an onset on or after dosing of MMF on run-in Day 1 up to the first double-blind dose, or any pre-existing condition that worsened. AE: any untoward medical occurrence that does not necessarily have a causal relationship with this treatment. SAE: any untoward medical occurrence that at any dose: results in death; in the view of the Investigator, places the participant at immediate risk of death (a life-threatening event); requires inpatient hospitalization or prolongation of existing hospitalization; results in persistent or significant disability/incapacity; or results in a congenital anomaly/birth defect. An SAE may also be any other medically important event that, in the opinion of the Investigator, may jeopardize the participant or may require intervention to prevent one of the other outcomes listed above.
Time Frame: Day 1 to Week 12
Population: All enrolled participants
Measure: Number; unit: participants
Groups:
- Run-In: All Enrolled Participants: At Run-in Day 1, participants entering the study received oral corticosteroid (prednisone or equivalent) starting at 0.75 mg/kg/day (maximum allowed dose of 60 mg/day) for 2 weeks and subsequently tapered over an 8-week period to 10 mg/day by Run-in Week 10. Following confirmation of eligibility, subjects also received MMF starting at Run-in Day 1 at a total dose of 1 g/day and titrated to a target dose of 2 g/day by Run-in Week 2.
Arm/Group | Run-In: All Enrolled Participants
Number analyzed (Participants) | 276
participants
  Any Event | 209
  Moderate or Severe Event | 94
  Severe Event | 18
  Related Event to MMF | 90
  Serious Event | 28
  Related Serious Event to MMF | 12
  Fatal Event | 2
  Discontinued Treatment Due to Event | 0
  Withdrew From Study Due to Event | 10

8. Secondary Outcome: Number of Participants With AEs, SAEs and AEs Leading to Study Discontinuation During the Double-Blind Period
Description: AEs that had an onset on or after dosing of BIIB023 or placebo, or any pre-existing condition that worsened. AE: any untoward medical occurrence that does not necessarily have a causal relationship with this treatment. SAE: any untoward medical occurrence that at any dose: results in death; in the view of the Investigator, places the participant at immediate risk of death (a life-threatening event); requires inpatient hospitalization or prolongation of existing hospitalization; results in persistent or significant disability/incapacity; or results in a congenital anomaly/birth defect. An SAE may also be any other medically important event that, in the opinion of the Investigator, may jeopardize the participant or may require intervention to prevent one of the other outcomes listed above.
Time Frame: Week 12 to Week 56
Population: The safety population was defined as all subjects who received at least 1 dose of study treatment (including placebo or BIIB023).
Measure: Number; unit: participants
Arm/Group | Placebo | BIIB023 3 mg/kg | BIIB023 20 mg/kg
Number analyzed (Participants) | 63 | 63 | 62
participants
  Any event | 48 | 60 | 53
  Moderate or severe event | 26 | 32 | 22
  Severe event | 4 | 6 | 5
  Event related to double-blind treatment | 5 | 15 | 11
  Event related to MMF | 21 | 24 | 22
  Serious event | 7 | 11 | 10
  Serious event related to double-blind treatment | 3 | 3 | 2
  Serious event related to MMF | 6 | 4 | 3
  Fatal event | 1 | 0 | 0

9. Secondary Outcome: Duration of Renal Response in Participants Who Achieve Partial or Complete Renal Response at Any Time During the Study
Description: Number of days between first visit with response to last consecutive visit with partial or complete response. Complete renal response is defined as: (1) uPCR <0.5 mg/mg with ≥ 50% reduction of uPCR from Day 1 (Baseline) (from a 24 hour urine collection); and (2) eGFR within normal range. Partial renal response is defined as: (1) ≥ 50% reduction in uPCR from Day 1 (Baseline; from a 24-hour urine collection) and, (2) with one of the following: (a) uPCR of < 1.0 mg/mg if the Day 1 (Baseline) was ≤ 3.0 mg/mg, or, (b) uPCR < 3.0 mg/mg if the Day 1 (Baseline) ratio was > 3.0 mg/mg; and stabilization of renal function (eGFR + or - 25% of Day 1 [Baseline] or serum creatinine within normal range). Estimated from the Kaplan-Meier Curve.
Time Frame: up to Week 52
Population: The ITT population included all participants who were randomized and received at least 1 dose of study treatment (BIIB023 or placebo).
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Placebo | BIIB023 3 mg/kg | BIIB023 20 mg/kg
Number analyzed (Participants) | 48 | 39 | 40
days | 48.3 (83.23) | 45.6 (75.42) | 52.1 (106.72)
Statistical Analysis 1: Comparison: Placebo vs BIIB023 3 mg/kg; Test type: Superiority or Other; p = 0.863, Regression, Cox
Statistical Analysis 2: Comparison: Placebo vs BIIB023 20 mg/kg; Test type: Superiority or Other; p = 0.769, Regression, Cox
Statistical Analysis 3: Comparison: Placebo vs BIIB023 3 mg/kg; Test type: Superiority or Other; p = 0.907, ANCOVA
Statistical Analysis 4: Comparison: Placebo vs BIIB023 20 mg/kg; Test type: Superiority or Other; p = 0.996, ANCOVA

ADVERSE EVENTS:
Time Frame: AEs: Run-in Day 1 through Week 64 +/- 5 days. SAEs: Screening through Week 64 +/- 5 days.
Groups:
- Run-in Period: At Run-in Day 1, participants entering the study received oral corticosteroid (prednisone or equivalent) starting at 0.75 mg/kg/day (maximum allowed dose of 60 mg/day) for 2 weeks and subsequently tapered over an 8-week period to 10 mg/day by Run-in Week 10. Following confirmation of eligibility, subjects also received MMF starting at Run-in Day 1 at a total dose of 1 g/day and titrated to a target dose of 2 g/day by Run-in Week 2.
- Placebo: Placebo intravenous (IV) infusion on Day 1, Week 2, Week 4, Week 8, and every 4 weeks thereafter through Week 48, plus background therapy including oral steroids (prednisone or equivalent) and MMF.
Arm/Group | Run-in Period | Placebo | BIIB023 3 mg/kg | BIIB023 20 mg/kg
Serious Adverse Events (participants affected / at risk) | 28/276 | 7/63 | 11/63 | 10/62
Other Adverse Events (participants affected / at risk) | 134/276 | 33/63 | 46/63 | 43/62
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Run-in Period (N=276) | Placebo (N=63) | BIIB023 3 mg/kg (N=63) | BIIB023 20 mg/kg (N=62)
Anaemia (Blood and lymphatic system disorders) | 2 | 0 | 0 | 0
Leukopenia (Blood and lymphatic system disorders) | 1 | 0 | 0 | 0
Acute myocardial infarction (Cardiac disorders) | 0 | 1 | 0 | 0
Cardiac failure (Cardiac disorders) | 1 | 0 | 0 | 0
Congestive cardiomyopathy (Cardiac disorders) | 0 | 0 | 0 | 1
Cataract (Eye disorders) | 0 | 1 | 0 | 0
Diarrhoea (Gastrointestinal disorders) | 2 | 0 | 0 | 0
Faecaloma (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Food poisoning (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Intestinal obstruction (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Vomiting (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Oedema (General disorders) | 1 | 0 | 0 | 0
Oedema peripheral (General disorders) | 0 | 0 | 0 | 1
Pyrexia (General disorders) | 0 | 0 | 1 | 0
Drug-induced liver injury (Hepatobiliary disorders) | 0 | 0 | 0 | 1
Brain abscess (Infections and infestations) | 0 | 0 | 1 | 0
Cellulitis (Infections and infestations) | 1 | 0 | 0 | 0
Cytomegalovirus infection (Infections and infestations) | 0 | 0 | 1 | 0
Dysentery (Infections and infestations) | 0 | 1 | 0 | 0
Endocarditis (Infections and infestations) | 0 | 1 | 0 | 0
Gastroenteritis (Infections and infestations) | 0 | 0 | 3 | 2
Herpes zoster (Infections and infestations) | 4 | 0 | 0 | 0
Meningitis (Infections and infestations) | 1 | 0 | 0 | 0
Peritonitis (Infections and infestations) | 1 | 0 | 0 | 0
Pneumocystis jirovecii pneumonia (Infections and infestations) | 1 | 0 | 0 | 0
Pneumonia (Infections and infestations) | 2 | 0 | 1 | 2
Pneumonia cytomegaloviral (Infections and infestations) | 1 | 0 | 0 | 0
Pyelonephritis acute (Infections and infestations) | 0 | 0 | 1 | 0
Respiratory tract infection (Infections and infestations) | 1 | 0 | 0 | 0
Sepsis (Infections and infestations) | 0 | 1 | 0 | 0
Sinusitis (Infections and infestations) | 1 | 0 | 0 | 0
Upper respiratory tract infection (Infections and infestations) | 0 | 1 | 0 | 0
Urinary tract infection (Infections and infestations) | 1 | 0 | 0 | 0
Urosepsis (Infections and infestations) | 1 | 0 | 0 | 0
Viral infection (Infections and infestations) | 1 | 0 | 0 | 0
Infusion related reaction (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0
Blood creatinine increased (Investigations) | 0 | 0 | 1 | 0
Dehydration (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1
Hypokalaemia (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0
Systemic lupus erythematosus (Musculoskeletal and connective tissue disorders) | 1 | 1 | 0 | 0
B-cell lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0
Transient ischaemic attack (Nervous system disorders) | 1 | 0 | 0 | 0
Acute kidney injury (Renal and urinary disorders) | 0 | 0 | 1 | 0
Glomerulonephritis rapidly progressive (Renal and urinary disorders) | 1 | 0 | 0 | 1
Lupus nephritis (Renal and urinary disorders) | 2 | 0 | 3 | 2
Renal failure (Renal and urinary disorders) | 0 | 0 | 1 | 0
Renal impairment (Renal and urinary disorders) | 1 | 0 | 0 | 0
Pulmonary alveolar haemorrhage (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1
Pulmonary congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1
Rash (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0
Papilloma excision (Surgical and medical procedures) | 1 | 0 | 0 | 0
Hypotension (Vascular disorders) | 0 | 0 | 0 | 1
Thrombosis (Vascular disorders) | 0 | 0 | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Run-in Period (N=276) | Placebo (N=63) | BIIB023 3 mg/kg (N=63) | BIIB023 20 mg/kg (N=62)
Anaemia (Blood and lymphatic system disorders) | 7 | 4 | 4 | 7
Leukopenia (Blood and lymphatic system disorders) | 10 | 7 | 5 | 2
Neutropenia (Blood and lymphatic system disorders) | 3 | 4 | 5 | 0
Diarrhoea (Gastrointestinal disorders) | 31 | 2 | 2 | 8
Nausea (Gastrointestinal disorders) | 14 | 3 | 5 | 2
Oedema peripheral (General disorders) | 8 | 1 | 4 | 1
Bronchitis (Infections and infestations) | 10 | 1 | 3 | 7
Gastroenteritis (Infections and infestations) | 9 | 6 | 6 | 7
Influenza (Infections and infestations) | 4 | 2 | 1 | 4
Nasopharyngitis (Infections and infestations) | 13 | 3 | 5 | 5
Upper respiratory tract infection (Infections and infestations) | 21 | 7 | 13 | 6
Urinary tract infection (Infections and infestations) | 8 | 2 | 6 | 2
Hypokalaemia (Metabolism and nutrition disorders) | 11 | 1 | 6 | 3
Arthralgia (Musculoskeletal and connective tissue disorders) | 10 | 6 | 6 | 5
Dizziness (Nervous system disorders) | 3 | 1 | 4 | 3
Headache (Nervous system disorders) | 12 | 6 | 7 | 6
Proteinuria (Renal and urinary disorders) | 1 | 3 | 5 | 6
Alopecia (Skin and subcutaneous tissue disorders) | 8 | 1 | 5 | 3
Rash (Skin and subcutaneous tissue disorders) | 8 | 4 | 4 | 0
Hypertension (Vascular disorders) | 10 | 0 | 4 | 5

LIMITATIONS AND CAVEATS:
Study was terminated based on the review of results following the prespecified, blinded futility analysis, which did not demonstrate sufficient efficacy to warrant continuation of the study. Study was not terminated based on safety considerations.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Our agreement is subject to confidentiality but generally the PI can publish, for noncommercial purposes only, results and methods of the trial, but no other Sponsor Confidential Information. PI must give Sponsor no less than 60 days to review any manuscript for a proposed publication and must delay publication for up to an additional 90 days thereafter if Sponsor needs to file any patent application to protect any of Sponsor's intellectual property contained in the proposed publication.